CLINICAL TRIAL: NCT00113594
Title: Population Pharmacokinetic Study in Adolescent Patients With Schizophrenia or Bipolar I Disorder Treated With Olanzapine
Brief Title: Olanzapine Treated Adolescents With Schizophrenia or Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9483; F1D-MC-HGMF
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
The purpose of this study is to characterize olanzapine pharmacokinetics: the inter- and intra- subject variabilities of olanzapine pharmacokinetics; and the potential influence of patient factors such as age, weight, gender, origin, and smoking status on olanzapine pharmacokinetics in adolescents with schizophrenia or bipolar I disorder. This study will also assess the safety of olanzapine delivered orally.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 13 through 17 years of age (must not have reached their 18th birthday prior to Visit 1).
* Female patients must not be pregnant or nursing.
* Patient and patient's parent/authorized legal representative must have a level of understanding sufficient to perform all tests and examinations required by the protocol, and must have given informed consent.
* Patient must have a previously documented diagnosis of schizophrenia or bipolar I according to the DSM-IV-TR, and either confirmed previously by K-SADS-PL or be confirmed by K-SADS-PL at Visit 1.

Exclusion Criteria:

* Patients must not be experiencing acute, serious, or unstable medical conditions other than schizophrenia or bipolar I disorder.
* Patients are not allowed into the study if they currently meet the criteria for the depressed phase of bipolar disorder or are diagnosed with Bipolar II Disorder.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2005-06; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To characterize olanzapine pharmacokinetics
The inter- and intra-subject variabilities of olanzapine pharmacokinetics
The potential influence of patient factors such as age, weight, gender, origin, and smoking status on olanzapine pharmacokinetics in adolescents 13-17 years of age that have been diagnosed with schizophrenia or bipolar I disorder

SECONDARY OUTCOMES:
To assess the safety of olanzapine delivered orally by measuring adverse events, change in vital signs, weight, laboratory analytes, electrocardiogram (ECG), and severity of extrapyramidal symptoms
To assess the effect of olanzapine on overall symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cerritos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Poway, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Eagle, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Olean, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Portsmouth, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kirkland, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, West Allis, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Juan, Puerto Rico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Moscow, Russia

REFERENCES:
- [Derived] Kryzhanovskaya LA, Robertson-Plouch CK, Xu W, Carlson JL, Merida KM, Dittmann RW. The safety of olanzapine in adolescents with schizophrenia or bipolar I disorder: a pooled analysis of 4 clinical trials. J Clin Psychiatry. 2009 Feb;70(2):247-58. doi: 10.4088/jcp.08m03538. Epub 2009 Feb 10. PMID 19210948
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com